CLINICAL TRIAL: NCT00724815
Title: The Efficacy and Tolerability of NP101, a Sumatriptan Iontophoretic Transdermal Patch, in the Treatment of Acute Migraine: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: The Efficacy and Tolerability of NP101 Patch in the Treatment of Acute Migraine
Acronym: NP101-007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NuPathe Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROT-15-NP101-007
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan (Experimental): NP101 - sumatriptan iontophoretic transdermal patch
  Interventions: Drug: NP101 - Sumatriptan iontophoretic transdermal patch
- Placebo (Placebo Comparator): Placebo iontophoretic transdermal patch
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NP101 - Sumatriptan iontophoretic transdermal patch — Sumatriptan iontophoretic transdermal patch
  Other Names: Sumatriptan
  Arms: Sumatriptan
Drug: Placebo — NP101 Placebo iontophoretic transdermal patch
  Other Names: NP101 Placebo
  Arms: Placebo

SUMMARY:
This study was a randomized, parallel group, double-blind, placebo controlled design to compare the efficacy and tolerability of NP101 to a placebo iontophoretic transdermal patch. The primary objective of this study was to assess the proportion of subjects who were headache pain free at two hours after patch activation.

Key secondary objectives included:

1. The proportion of subjects who were nausea free at two hours after patch activation.
2. The proportion of subjects who were photophobia free at two hours after patch activation.
3. The proportion of subjects who were phonophobia free at two hours after patch activation.

DETAILED DESCRIPTION:
Subjects stayed in the study until they had treated one migraine headache with a study patch or two months after randomization, whichever occurred first. During a migraine headache, subjects rated their baseline headache pain severity in a Migraine Study Diary using a 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) and applied the study patch only if their score was 2 or 3 (i.e., qualifying migraine headache). In addition to headache pain severity, subjects also recorded the presence or absence of aura, nausea, phonophobia, and photophobia, as well as the location of their headache (unilateral or bilateral) and whether their headache increased with movement.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult male or female, age range 18 years to 65 years.
* Subject has a diagnosis of migraine headache, with or without aura, as defined in the ICDH-II and the diagnosis was made before the age of 50.
* Subject typically experiences moderate to severe headaches during a migraine attack.
* Subject has at least a one year history of migraine.
* Subject will be judged to be in good health, based on results of a medical history, physical examination, vital signs, ECG and laboratory profile.
* Female subject of childbearing potential must have a negative pregnancy test at screening and prior to randomization.
* Subject must have a negative drug screen.
* Subject must be capable of reading and understanding either English or Spanish subject information materials. Be able to successfully apply a practice patch, carry-out all subject procedures, and be able to voluntarily sign and date an IRB approved IC agreement.
* Subject has an acceptable patch application site (upper arm) that is relatively hair free and has no scars, tattoos, scratches, or bruises.

Exclusion Criteria:

* Subject has or plans to start, stop, or change treatment or dose with prophylactic anti-migraine treatment within 3 months prior to the subjects' study randomization date and through the final visit.
* Subject has or plans to start, stop, or change treatment or dose of any of the following within 3 months prior to the subjects' study randomization date through final visit: anxiolytics, lithium and other mood stabilizers, hypnotics or antipsychotics.
* Subject had less than one migraine per month or more than six migraines per month, or more than 15 headache days per month for any of the three months prior to randomization.
* Subject has suspected or confirmed cardiovascular disease that contraindicates study participation.
* Subject has a history of epilepsy or conditions associated with a lowered seizure threshold.
* Subject has Raynaud's disease.
* Subject has a history of basilar or hemiplegic migraines.
* Subject has a current diagnosis of a major depressive disorder per the DSM IV R.
* Subject has a history (within 1 year) or current evidence of drug or alcohol abuse or dependence.
* Subject is unwilling to discontinue use of serotonin agonists (triptans), except for the study patch, through the Final Visit.
* Subject has taken SSRI's, SNRI's, TCA's, MAOI's or preparations containing St. John's Wort within 1 month prior to screening and/or is planning to start any of these medications during the study.
* Subject is unwilling to discontinue use of a PD-5 inhibitors through the Final Visit.
* Subject has taken ergot medications within 7 days prior to Randomization and/or is unwilling to discontinue use through the Final Visit.
* Subject has a history of a significant allergy or hypersensitivity to any component of the study patch.
* Subject has any generalized skin irritation or disease including eczema, psoriasis, melanoma, or contact dermatitis.
* Subject has clinically significant abnormal laboratory parameters, vital signs or ECG parameters.
* Subject is known to be hepatitis B, hepatitis C or HIV positive.
* Subject has hepatic dysfunction based on laboratory results or if in the opinion of the Investigator the subject's history, physical examination or other laboratory tests suggest hepatic dysfunction.
* Female subject who is pregnant, breast feeding, or if of childbearing potential, is not using or is unwilling to use an effective form of contraception during the study and for a period of 30 days following dosing.
* Subject has known history of failure to respond to sumatriptan.
* Subject has participated in a clinical study within 30 days of screening or is planning to participate in another clinical study.
* Subject has been previously enrolled in NP101-007
* Subject is electrically sensitive or who have electrically sensitive support systems (e.g., pacemaker).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pierce, MD, Study Director — NuPathe Inc.
Locations (34):
- United States (34):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Newport Beach, California
  - San Francisco, California
  - Santa Monica, California
  - Fairfield, Connecticut
  - Ocala, Florida
  - Palm Beach Gardens, Florida
  - Sunrise, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Decatur, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Springfield, Missouri
  - St Louis, Missouri
  - Mount Vernon, New York
  - Plainview, New York
  - Greensboro, North Carolina
  - West Chester, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wynnewood, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Alexandria, Virginia
  - Virginia Beach, Virginia
  - Seattle, Washington

REFERENCES:
- [Derived] Goldstein J, Smith TR, Pugach N, Griesser J, Sebree T, Pierce M. A sumatriptan iontophoretic transdermal system for the acute treatment of migraine. Headache. 2012 Oct;52(9):1402-10. doi: 10.1111/j.1526-4610.2012.02198.x. Epub 2012 Jun 13. PMID 22694484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated January 2009 and completed July 2009. Patients were enrolled from 38 investigative sites across the United States.
Groups:
- NP101 Patch: The NP101 patch contained 86 mg of sumatriptan and was designed to deliver approximately 6.5 mg of sumatriptan over 4 hours. Patients were asked to treat one migraine episode with moderate to severe headache pain.
- Placebo Patch: The study placebo patch contained sodium chloride instead of sumatriptan which was delivered over 4 hours. Patients were asked to treat one migraine episode with moderate to severe headache pain.
Period: Overall Study
Arm/Group | NP101 Patch | Placebo Patch
Started | 265 (subjects randomized) | 265 (subjects randomized)
Completed | 222 | 226
Not Completed | 43 | 39
Not completed — Randomized, not treated | 31 | 30
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Other Various | 3 | 5

BASELINE CHARACTERISTICS:
Population: Per protocol, the safety population was defined as subjects who applied a study patch. In each treatment group there were subjects who were randomized but not treated (NP101=31, placebo patch=30) and are therefore not included in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | NP101 Patch | Placebo Patch | Total
Number analyzed (Participants) | 234 | 235 | 469
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 233 | 235 | 468
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (11.20) | 41.2 (11.06) | 40.8 (11.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 201 | 398
  Male | 37 | 34 | 71
Region of Enrollment [Number; unit: participants]
  United States | 234 | 235 | 469

OUTCOME MEASURES:

1. Primary Outcome: Pain Free at Two Hours
Description: Subjects whose headache severity score equaled zero (0) two hours post patch activation and who had not received any rescue medication before their two-hour assessment.
Time Frame: 2 hours post patch activation
Population: Per protocol, the intent-to-treat population was assessed.
Measure: Number; unit: participants
Arm/Group | NP101 Patch | Placebo Patch
Number analyzed (Participants) | 226 | 228
participants | 40 [1.2 to 3.7] | 21 [1.2 to 3.7]

2. Secondary Outcome: Photophobia Free at Two Hours
Description: Subjects who were photophobia free and who had not received any rescue medication before their two-hour assessment.
Time Frame: 2 hours post patch activation
Population: Per protocol, the intent-to-treat population was assessed.
Measure: Number; unit: participants
Arm/Group | NP101 Patch | Placebo Patch
Number analyzed (Participants) | 226 | 228
participants | 116 | 83

3. Secondary Outcome: Phonophobia Free at Two Hours
Description: Subjects who were phonophobia free and who had not received any rescue medication before their two-hour assessment.
Time Frame: 2 hours post patch activation
Population: Per protocol, the intent-to-treat population was assessed.
Measure: Number; unit: participants
Arm/Group | NP101 Patch | Placebo Patch
Number analyzed (Participants) | 226 | 228
participants | 125 | 89

4. Secondary Outcome: Nausea Free at Two Hours
Description: Number of subjects who were nausea free and who had not received any rescue medication before their two-hour assessment.
Time Frame: 2 hours post patch activation
Population: Per protocol, the intent-to-treat population was assessed.
Measure: Number; unit: participants
Arm/Group | NP101 Patch | Placebo Patch
Number analyzed (Participants) | 226 | 228
participants | 189 | 144

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from study screening until 30 days post patch removal.
Arm/Group | NP101 Patch | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 0/234 | 0/235
Other Adverse Events (participants affected / at risk) | 114/234 | 100/235
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NP101 Patch (N=234) | Placebo Patch (N=235)
Application site pain (General disorders) | 54 (54) | 34 (34)
Application site paraesthesia (General disorders) | 28 (28) | 44 (44)
Application site pruritus (General disorders) | 18 (18) | 16 (16)
Application site reaction (General disorders) | 16 (16) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the study agreement, Investigators have the right to publish or present information and/or data arising from the study, provided the text of any such publication or presentation is submitted for review at least thirty days prior to submission for publication or other disclosure and NuPathe shall have the right to request the removal of any confidential information.